CLINICAL TRIAL: NCT07242664
Title: A Trial to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Insulin GZR33 Compared With Insulin Degludec at Steady State in Participants With Type 1 Diabetes
Brief Title: Clamp Study to Estimate the Relative Potency of GZR33 Versus Insulin Degludec at Steady State
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GZR33-T1D-US101
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes Mellitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1 - GZR-33, period 2 insulin degludec (Experimental): Period 1 - GZR-33 once daily for six days. Post wash-out, insulin degludec once daily for six days
  Interventions: Drug: GZR-33
- Period 1 - insulin degludec, period 2 - GZR-33 (Experimental): Period 1 - insulin degludec once daily for six days. Post wash-out, GZR-33 once daily for six days
  Interventions: Drug: GZR-33

INTERVENTIONS:
Drug: GZR-33 — GZR33 is a long-acting basal insulin analogue

SUMMARY:
This trial intends to investigate the pharmacodynamics, pharmacokinetics, safety, and tolerability of insulin GZR33 (hereafter referred to as GZR33) and estimate its potency in comparison with insulin degludec.

ELIGIBILITY:
Inclusion Criteria: type 1 diabetes for at least 12 months

* 18-64 years of age
* HbA1c <= 9.0%.
* Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2
* treated with a stable insulin regimen for at least 2 months, in a dose > 0.2 and < 1.2 U/kg/day

Exclusion Criteria:

* blood pressure outside the range 90 to 140 mmHg (systolic) or 50 to 99 mmHg (diastolic)
* clinically significant concomitant diseases
* recurrent severe hypoglycemia (more than 1 severe hypoglycemic episode requiring assistance from another person within 180 days before screening)
* hypoglycemia unawareness
* estimated glomerular filtration rate (eGFR) <60.0 mL/min/1.73 m2

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
the relative potency of GZR33 to insulin degludec | a two week run-in phase
  Primary endpoint will be the relative potency of GZR33 to insulin degludec, according to the following equation:
  Relative Potency = GIR24h,ss,GZR33 /GIR24h,ss,degludec) × (Dosedegludec/DoseGZR33).

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Profil Institut, Neuss
  - Profil, Neuss